CLINICAL TRIAL: NCT02785796
Title: Effects of Cranial Manipulation in Healthy Patients Revealed by Salivary Alpha Amylase Activity
Brief Title: Effect of Cranial Manipulation on ANS Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Accademia Italiana Medicina Osteopatica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 001
Record Dates: First submitted 2016-05-19; First posted 2016-05-30 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Alpha Amylase; Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- CV4 (Experimental): The practitioner will contact the participant's occiput (lateral to the external occipital protuberances, but medial to the occipital-mastoid suture) with his or her thenar eminences. When no cranial mobility will be found, operators will be free to use any kind of technique to enhance the cranial movement before CV4 procedure. Once the practitioner will detect the CRI, the practitioner will resist the flexion phase of the CRI and exaggerate the extension phase. This compressive pressure will be maintained until the CRI stopped, and the still-point is reached. The still-point will be held until the CRI return, at which point the compressive pressure will be slowly release
  Interventions: Other: CV4
- sham technique (Placebo Comparator): The operator will overlap the hands so that the thumbs formed a "V". The operator's thenar eminences will contact the occiput very lightly well below the positioning used in the CV4 procedure but with no pressure on the occiput between the occipitomastoid sutures. Once placement will be achieved, the operator's hands will remain motionless for 10 min. Finally, the practitioner's hands will be gently removed and the participant's head will be placed on the table for both procedures
  Interventions: Other: SHAM TECHNIQUE
- Control (No Intervention): The control group will not receive ant type of treatment: subject just stay quietly in supine position in ambulatory room for ten minutes

INTERVENTIONS:
Other: CV4
  Arms: CV4
Other: SHAM TECHNIQUE
  Arms: sham technique

SUMMARY:
In osteopathy is generally believed that the cranial bones are equipped with an inherent mobility, which like any other joint may face restrictions on movement and then somatic dysfunction. For this reason, different techniques are used with the aim of increasing the mobility of the cranial bones. Some of these have been effective in modifying physiological parameters related to the activity of the autonomic nervous system, such as cardiac function or sleep latency. This study aims to test the effectiveness of a specific craniosacral technique, compression of the fourth ventricle CV4, using the salivary marker alpha amylase, which is sensitive to changes in the activity of the autonomic nervous system. To patients recruited from students of AIMO, we will ask to provide saliva samples before and after CV4 treatment. In particular, saliva will be collected four times per patient: at the initial time, after administration of a stressful event (hand immersion in ice water), immediately after application of the CV4 technique and thirty minutes after the application of the CV4 technique. For each sample of saliva detected, we will proceed to measure the activity of alpha amylase and flow rate, variables sensitive to the activation of the autonomic nervous system.

DETAILED DESCRIPTION:
A minimum of 90 healthy subjects ranging from 20 to 25 years will be selected from students in Accademia Itliana di Medicina Osteopatica, Saronno, Italy (AIMO) and randomly assigned to the placebo, control or the CV4 arm. Randomization will account for sex and score in the STAI- 2 (form Y) questionnaire, assessing trait anxiety for each subject.

Every sampling session will be taken from 10.00 AM to 1.00 PM to minimize the effect of diurnal variation in salivary alpha-amylase activity. Subjects will be instructed to abstain from eating, smoking, drinking any beverages and exercising 2h before the experiment because these activities has been shown to have an influence on sAA activity.

The day of treatment each subject will completed the STAI-1 (form Y) questionnaire to evaluate the anxiety of the moment. Saliva collection will be made by passive drooling continuously for 5 minutes in a 15 ml falcon tube. Saliva will be collected before, immediately after and 30 minutes after application of a true CV4 technique or application of a sham technique performed by different osteopaths. Saliva samples will be immediately frozen at -20°C for subsequent analysis.

Operators will be osteopaths trained in cranial field. The application of the CV4 and sham protocols will occur in an examination room setting. The subject will lie in supine position with the operator at the head of the treatment table with forearms resting on table either for CV4 either for the sham procedure.

For the CV4 technique the practitioner will contact the participant's occiput (lateral to the external occipital protuberances, but medial to the occipital-mastoid suture) with his or her thenar eminences. When no cranial mobility will be found, operators will be free to use any kind of technique to enhance the cranial movement before CV4 procedure. Once the practitioner will detect the CRI, the practitioner will resist the flexion phase of the CRI and exaggerate the extension phase. This compressive pressure will be maintained until the CRI stopped, and the still-point is reached. The still-point will be held until the CRI return, at which point the compressive pressure will be slowly release. For the sham CV-4, The operator will overlap the hands so that the thumbs formed a "V". The operator's thenar eminences will contact the occiput very lightly well below the positioning used in the CV4 procedure but with no pressure on the occiput between the occipitomastoid sutures. Once placement will be achieved, the operator's hands will remain motionless for 10 min. Finally, the practitioner's hands will be gently removed and the participant's head will be placed on the table for both procedures.

Flow rate will be measured for samples thawed by 5 ml graduated capillary. Samples will be then centrifuged (for ten minutes at 3000 rpm) and the supernatant collect in clean Eppendorf tubes. Salivary alpha-amylase activity will be then measured by a commercial kit (IBL) and a spectrophotometer for the optical reading.

ELIGIBILITY:
Inclusion Criteria:

* consensus signed

Exclusion Criteria:

* oral contraceptive
* drugs assumption
* pathology of oral cavity
* failure to comply the directives

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-05; Primary Completion 2016-05 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
alpha amylase activity measured by enzymatic assay | measurement before the technique application
salivary flow rate | measurement before the technique application
alpha amylase activity measured by enzymatic assay | measurement immediately after the technique application
alpha amylase activity measured by enzymatic assay | measurement 30 minutes after the technique application
salivary flow rate | measurement immediately after the technique application
salivary flow rate | measurement 30 minutes after the technique application

CONTACTS AND LOCATIONS:
Locations (1):
- AIMO, Saronno, Varese, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cutler MJ, Holland BS, Stupski BA, Gamber RG, Smith ML. Cranial manipulation can alter sleep latency and sympathetic nerve activity in humans: a pilot study. J Altern Complement Med. 2005 Feb;11(1):103-8. doi: 10.1089/acm.2005.11.103. PMID 15750368
- [Background] Nater UM, Rohleder N. Salivary alpha-amylase as a non-invasive biomarker for the sympathetic nervous system: current state of research. Psychoneuroendocrinology. 2009 May;34(4):486-96. doi: 10.1016/j.psyneuen.2009.01.014. Epub 2009 Feb 26. PMID 19249160